CLINICAL TRIAL: NCT02156674
Title: Study of Administration of Intravenous Naglazyme® Following Allogeneic Transplantation for Maroteaux-Lamy Syndrome
Brief Title: Naglazyme After Allo Transplant for Maroteaux-Lamy Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014LS014; MT2014-08R (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Maroteaux-Lamy Syndrome
Keywords: Maroteaux-Lamy Syndrome; mucopolysaccharide VI; MPS VI
MeSH Terms: conditions — Mucopolysaccharidosis VI | interventions — galsulfase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naglazyme® (Experimental): weekly Naglazyme® infusion for 2 years
  Interventions: Drug: Naglazyme®

INTERVENTIONS:
Drug: Naglazyme® — 1 mg per kg of body weight administered once weekly as an intravenous infusion

SUMMARY:
This is a single center study in which Naglazyme® will be given weekly for two years in patients with Maroteaux-Lamy syndrome, also known as mucopolysaccharide VI (MPS VI), who have previously been treated with an allogeneic transplant.

ELIGIBILITY:
Inclusion Criteria:

* Mucopolysaccharidosis type VI (MPS VI, Maroteaux-Lamy syndrome) treated with a prior allogeneic transplant >2 years previously
* Persons currently receiving Naglazyme may be accepted into the study
* Age > 2 years
* >10% engrafted based on most recent testing
* Willing to commit to traveling to the University of Minnesota every 6 months
* Written informed consent with parent/guardian consent for children < 18 years of age or persons unable to consent with minor assent if appropriate

Exclusion Criteria:

* History of cardiac or pulmonary insufficiency or those requiring continuous supplemental oxygen
* Pregnant or breastfeeding
* Any condition that, in the view of the investigator, places the patient at high risk of poor treatment compliance or of not completing the study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Braulin, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naglazyme®
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Naglazyme®
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Glycosaminoglycan (GAG) Excretion
Description: Change in urinary glycosaminoglycan (GAG) excretion from baseline to 2 years
Time Frame: Baseline and 2 years
Measure: Number; unit: mg/mm Cr
Arm/Group | Naglazyme®
Number analyzed (Participants) | 1
mg/mm Cr | -0.8

2. Primary Outcome: Change in Distance Traveled
Description: Change in distance traveled in 6 minute walk and standard tests of range of motion and mobility. Improvement in distance walked from the start to study to end of the study is reported
Time Frame: Baseline and 2 years
Measure: Number; unit: Foot
Arm/Group | Naglazyme®
Number analyzed (Participants) | 1
Foot | 136

3. Primary Outcome: Change in Neurocognitive Ability
Description: Subjects will undergo full neuropsychological testing annually and abbreviated testing for attention and adaptive skills at the six-month interval visits
Time Frame: Baseline and 2 years
Population: Not Evaluated
Arm/Group | Naglazyme®
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Development of Neutralizing Antibodies to Naglazyme Therapy
Description: Development of antibodies including neutralizing antibodies with weekly Naglazyme therapy and the impact of these antibodies on cardiorespiratory and skeletal parameters as measured by the 6--minute walk test and standard tests of range of motion and mobility, and the change in neurocognitive ability.
  Anti-rhASB antibodies in patient's sera were tested in the Biomarin Laboratory using an in-house test of ELISA.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Naglazyme®
Number analyzed (Participants) | 1
participants | 0

5. Secondary Outcome: Number of Participants With Development of Neutralizing Antibodies to Naglazyme Therapy
Description: as for outcome 4
Time Frame: 2 years
Population: No data available
Arm/Group | Naglazyme®
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Naglazyme®
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT02156674/Prot_SAP_000.pdf